CLINICAL TRIAL: NCT02809690
Title: Pilot Feasibility Study of 18F-FMAU PET for Diagnosing and Characterizing Prostate Cancer
Brief Title: 18F-FMAU PET/CT in Diagnosing and Characterizing Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4P-16-3; NCI-2016-00814 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 4P-16-3 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH); R21EB017568 (NIH)
Record Dates: First submitted 2016-06-19; First posted 2016-06-22 (Estimated); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Prostate Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Tomography, X-Ray Computed; Tomography; clevudine; Positron-Emission Tomography; Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (18F-FMAU PET/CT) (Experimental): Patients receive radiotracer F 18 d-FMAU IV over 1 minute and then undergo 18F-FMAU PET/CT on day 1. Patients then undergo standard of care multiparametic MRI and standard of care transrectal ultrasound-guided biopsy.
  Interventions: Device: CAT; Drug: 18F-FMAU; Other: Laboratory Biomarker Analysis; Procedure: Multiparametric Magnetic Resonance Imaging; Device: Positron Emission Tomography; Device: Ultrasound

INTERVENTIONS:
Device: CAT — Undergo 18F-FMAU PET/CT
  Other Names: CAT Scan; Computed Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT SCAN; tomography
Drug: 18F-FMAU — Patients receive radiotracer F 18 d-FMAU IV over 1 minute and then undergo 18F-FMAU PET/CT
  Other Names: Fluorine F 18 d-FMAU; 2'-deoxy-2'-[18F]fluoro-5-methyl-1-beta-D-arabinofuranosyluracil
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Multiparametric Magnetic Resonance Imaging — Undergo mpMRI
  Other Names: Multiparametric MRI
Device: Positron Emission Tomography — Undergo 18F-FMAU PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Device: Ultrasound — Undergo TRUS-guided biopsy

SUMMARY:
This pilot clinical trial studies how well fluorine F 18 d-FMAU (18F-FMAU) positron emission tomography (PET)/computed tomography (CT) works in diagnosing and characterizing prostate cancer. A PET/CT scan is an imaging test that uses a small amount of radioactive tracer that is given through the vein to take detailed pictures of areas inside the body where the tracer is taken up. Radiotracers such as 18F-FMAU may help to find the cancer and see how far the disease has spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To perform a prospective clinical imaging evaluation of 18F-FMAU PET/CT in addition to multiparametric magnetic resonance imaging (mpMRI) and standard transrectal ultrasound (TRUS)-guided 12-core biopsy for detection and localization of primary tumor in 40 men with suspected prostate cancer based on elevated/rising prostate specific antigen level, abnormal digital rectal exam, or those with prior negative standard biopsy who are now returning for a standard of care follow-up.

II. To examine the associations between the PET derived imaging parameters, serum PSA, mpMRI parameters (apparent diffusion coefficient [ADC], Ktrans) and the biopsy histopathology parameters.

OUTLINE:

Patients receive radiotracer F 18 d-FMAU intravenously (IV) over 1 minute and then undergo 18F-FMAU PET/CT on day 1. Patients then undergo standard of care multiparametic MRI and standard of care transrectal ultrasound-guided biopsy.

After completion of study treatment, patients are followed up at 24-96 hours.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo standard of care biopsy for suspected prostate cancer, or re-biopsy with prior negative systemic biopsy or restaging biopsy in patients with known prostate cancer on active surveillance

Exclusion Criteria:

* History of myocardial infarction within 6 months of the enrollment
* Active infection (except mild upper respiratory infections)
* Active prostatitis
* Non-prostate cancers currently on treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Proportion of men for whom biopsy cores taken based only on the 18F-FMAU PET/CT results would have yielded the same overall diagnosis as the standard TRUS-guided core or the mpMRI-directed prostate biopsies | Up to 1 year
  Standard descriptive methods will be used to summarize the data collected: means, standard deviations, ranges, and confidence intervals (or medians, quartiles), contingency tables, histograms, correlation coefficients (Pearson or Spearman) and scatter plots. The scatter plots and correlations between each of the histopathology parameters and the imaging parameters will be examined to better understand the relationships.
Proportion of men for whom the 18F-FMAU PET/CT identified all lesions that were found to have cancer based on the standard TRUS-guided and the mpMRI directed core prostate biopsies | Up to 1 year
  Standard descriptive methods will be used to summarize the data collected: means, standard deviations, ranges, and confidence intervals (or medians, quartiles), contingency tables, histograms, correlation coefficients (Pearson or Spearman) and scatter plots. The scatter plots and correlations between each of the histopathology parameters and the imaging parameters will be examined to better understand the relationships.
Proportion of men who completed both imaging procedures and for whom biopsy cores taken based only on the fluorine 18F-FMAU PET/CT results would have yielded the same overall diagnosis as the standard TRUS-guided core prostate biopsies | Up to 1 year
  Standard descriptive methods will be used to summarize the data collected: means, standard deviations, ranges, and confidence intervals (or medians, quartiles), contingency tables, histograms, correlation coefficients (Pearson or Spearman) and scatter plots. The scatter plots and correlations between each of the histopathology parameters and the imaging parameters will be examined to better understand the relationships.

CONTACTS AND LOCATIONS:
Overall Officials: Hossein Jadvar, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States